CLINICAL TRIAL: NCT03368820
Title: Cardiovascular Morbidities and Lung Cancer Treatment
Brief Title: Cardiovascular Morbidities and Lung Cancer Treatment: a Prospective Registry
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: European Lung Cancer Working Party (Other)
Responsible Party: Sponsor
Other Study IDs: 01151
Record Dates: First submitted 2017-11-24; First posted 2017-12-11 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Lung Neoplasm
Keywords: lung neoplasms; cardiovascular co-morbidity
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — Treatment left at the discretion of the participant

SUMMARY:
Therapeutic algorithms for lung cancer are mainly based on randomised controlled trials which excluded patients with severe co-morbidities. Smoking, the main risk factor for lung cancer, is associated with cardiovascular events that may impact on the therapeutic decision.

The aim of this registry is to determine if and how cardiovascular co-morbidities impact on the physicians' decision for anticancer treatment in lung cancer patients by comparing it to the European Lung Cancer Working Party (ELCWP) guidelines

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of lung cancer, either NSCLC or SCLC patients and carcinoid tumours
* Untreated lung cancer of any stage and any treatment (including palliative care only).
* Availability for participating in the detailed follow-up of the protocol.
* Signed informed consent.
* Age above 18 years.
* Presence of at least one co-morbidity:
* Any active or past cardiac ischemia
* Reduced left ventricular ejection fraction (< 50%)
* Obstructive cardiomyopathy
* Valvular dysfunction (3 or 4/4; valvular replacement)
* Arrhythmia (atrial flutter or fibrillation, significant ventricular arrhythmia, 2nd-3rd degree auriculo-ventricular block, Wolf-Parkinson-White and other similar aberrant conduction, bifascicular block, arrhythmogenic right ventricular dysplasia)
* Uncontrolled hypertension (systolic blood pressure (BP) > 160 millimeter of mercury (mmHg) or diastolic BP > 100 mmHg on ≥ 1 hypotensive drug) or controlled hypertension on ≥ 2 concurrent hypotensive drugs
* Active or treated peripheral arteritis (grade 2 or more)
* Cerebrovascular events
* Pulmonary embolism and/or thrombophlebitis or patients at high risk of thrombophilia (homozygous Leiden factor…)
* Aortic aneurism

Exclusion Criteria:

* Thymoma and thymic malignancies, pleural mesothelioma.
* Patient previously treated for lung cancer.
* Tumours for which complete staging cannot be assessed.
* History of prior malignant tumour, except non-melanoma skin cancer or in situ carcinoma of the cervix or of the bladder or cured malignant tumour (more than 5-year disease free interval).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any untreated lung cancer whatever the treatment intent
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-12-04 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Treatment decision adequacy | 1 year
  Comparison of physician's treatment decision to current ELCWP guidelines

SECONDARY OUTCOMES:
Treatment decision adequacy according to histology | 1 year
  Comparison of physician's treatment decision to current ELCWP guidelines separately in small (SCLC) and non-small lung cancer (NSCLC)
Response rate | Every 3 cycles for chemotherapy (9 weeks) or 1 month after completion of radiochemotherapy (15 weeks)
  Response rate in patients with cardiovascular co-morbidities and adapted treatment using (World Health Organisation (WHO) criteria
Overall survival | 1 year
  Survival will be measured from the day of diagnostic biopsy. All patients have to be followed until death

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Berghmans, MD, PhD, Study Chair — ELCWP
Locations (6):
- Belgium (6):
  - Department of Intensive Care Unit and Thoracic Oncology Institut Jules Bordet, Brussels
  - Hôpital Saint-Joseph, Charleroi
  - CHU Tivoli, La Louvière
  - Hôpital Ambroise Paré, Mons
  - CH Peltzer-La Tourelle, Verviers
  - Hôpital Mont-Godinne, Yvoir

IPD SHARING:
Plan to Share IPD: No